## Statistical analysis

A descriptive analysis of the variables included was carried out, where the quantitative variables are expressed as mean and standard deviation, and median with their respective ranges. Categorical variables are described based on their absolute number and percentage.

For the comparative analysis of the quantitative variables between admission and discharge, the Wilcoxon test for paired samples was used.

In the comparative analysis of the three variables evaluated between discharge, 3, 6 and 12 months, a comparison was made using the nonparametric Friedman test and a sensitivity analysis was performed with the Quade test. For the comparison between the different groups, the Nemenyi test was used. The missing data were imputed with the last registered value, in case of death the value with 0 was imputed.